CLINICAL TRIAL: NCT01731639
Title: The Influence of Motile Sperm Organelle Morphology Examination on ICSI Outcomes
Brief Title: Motile Sperm Organelle Morphology Examination (MSOME) Influence on Intracytoplasmic Sperm Injection (ICSI) Outcomes in Infertile Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sapientiae Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: MSOME_Grades
Record Dates: First submitted 2012-11-12; First posted 2012-11-22 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSOME (Experimental): The samples will be evaluated under high magnification
  Interventions: Other: MSOME

INTERVENTIONS:
Other: MSOME — The semen samples will be evaluated according to the 2010 WHO reference values. After ICSI 200 spermatozoa of each sample will be analyzed under high magnification (MSOME - x6600) and graded into four groups according to the presence or size of the vacuoles. Grade I: normal form and no vacuoles; grade II: normal form and ≤ 2 small vacuoles; grade III: normal form > 2 small vacuoles or at least one large vacuole and grade IV: large vacuole and abnormal head shapes or other abnormalities.

SUMMARY:
A new technique based on the motile sperm organelle morphology examination (MSOME) at a magnification of at least ×6000 has been developed. The MSOME assesses the nucleus, for both shape and chromatin content, which is the most important sperm organelle in influencing intracytoplasmic sperm injection (ICSI) outcomes.

DETAILED DESCRIPTION:
Sperm morphology has been described as one of the major determinants of male in vitro fertility. However, the standard morphology evaluation on random stained cells from the ejaculate is of limited value during ICSI. Current research is directed towards the dysmorphisms of the sperm head.A new technique based on the motile sperm organelle morphology examination (MSOME) at a magnification of at least ×6000 has been developed. The MSOME assesses the nucleus, for both shape and chromatin content, which is the most important sperm organelle in influencing ICSI outcomes. The goals for this study are to identify whether there is a connection between morphologic sperm normalcy under high magnification and (i) semen analysis according to the new World Health Organization (WHO) reference values and (ii) ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing ICSI as result of male factor or tubal factor or unexplained infertility
* Women with regular menstrual cycles of 25-35 days
* Women with normal basal follicle stimulating hormone (FSH) and luteinizing hormone (LH) levels
* Women with body mass index (BMI) less than 30 kg/m2
* Women with both ovaries and intact uterus

Exclusion Criteria:

* Women with polycystic ovaries syndrome
* Women with endometriosis
* Women with gynaecological/medical disorders
* Couples with any sexually transmitted disease
* Women who had received any hormone therapy for less than 60 days preceding the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates | 1 month
  Number of clinical pregnancy rate divided by the number of couples in which embryo transfer was performed.

SECONDARY OUTCOMES:
Implantation rates | 1 month
  Number of gestational sacs divided by the number of transferred embryos.

CONTACTS AND LOCATIONS:
Overall Officials: Edson Borges Jr., MD., PhD, Principal Investigator — Sapientiae Institute
Locations (1):
- Sapientiae Institute, São Paulo, São Paulo, Brazil